CLINICAL TRIAL: NCT03984175
Title: Implementation of Computerized Clinical Decision Support for Mechanical Ventilation of Patients With Acute Respiratory Distress Syndrome
Brief Title: Clinical Decision Support for Mechanical Ventilation of Patients With ARDS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: National Institutes of Health (NIH) (NIH); McKay-Dee Hospital (Other); Utah Valley Hospital (Unknown); Dixie Regional Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1050867
Record Dates: First submitted 2019-06-03; First posted 2019-06-12 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: ARDS; Lung Protective Mechanical Ventilation; Clinical Decision Support
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: Before and After Comparison
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with ARDS at three Intermountain tertiary hospitals (Experimental)
  Interventions: Procedure: Implementation of Processes

INTERVENTIONS:
Procedure: Implementation of Processes — Implementation of processes to improve compliance with low tidal volume ventilation in patients with ARDS using a computerized protocol

SUMMARY:
Perform a pilot study of quality improvement interventions for critical care physicians (intensivists) and respiratory therapists (RTs) to improve application of low tidal volume mechanical ventilation (LTVV) for patients with the acute respiratory distress syndrome (ARDS) using the computerized mechanical ventilation protocols currently available in the investigator's Cerner electronic health record (EHR).

DETAILED DESCRIPTION:
A multidisciplinary team of implementation researchers and clinical effectiveness researchers has been assembled to adapt the Consolidated Framework for Implementation Research (CFIR) for this planning study. The team identified the baseline clinical care delivery for LTVV in patients with ARDS across Intermountain hospitals and identified the barriers and facilitators to this standard of care. This pilot implementation study will focus on a Pilot Solution aimed at achieving ideal clinical care delivery of LTVV for patients with ARDS.

Abbreviations for Mechanical Ventilation:

PEEP: positive end expiratory pressure FIO2: fraction of inspired oxygen CPAP: continuous positive airway pressure PS: pressure support VC: volume control VC+: hybrid mode for volume targeted ventilation on Puritan Bennett ventilators PRVC: pressure regulated volume control, hybrid mode for volume targeted ventilation on Draeger ventilators PF ratio: ratio of partial pressure of arterial oxygen (PaO2 mmHg) divided by the FIO2 expressed in liters

ELIGIBILITY:
Inclusion Criteria:

1. Invasive mechanical ventilation
2. PF ratio <255
3. Bilateral infiltrates on chest radiograph (adjudicated by a co-investigator)
4. Presence of ≥1 risk factor for ARDS as determined by review of the HER

Exclusion Criteria:

1. Age <18 years
2. Pulmonary capillary wedge pressure >18 mm Hg if a right heart catheter is present
3. Prisoner
4. Known to be pregnant
5. Death <24 hours from initial intubation
6. Placed comfort care <24 hours from initial intubation
7. Mechanically ventilated for >7 days prior to meeting ARDS criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2018-07-08 (Actual); Primary Completion 2022-12-23 (Estimated); Study Completion 2022-12-23 (Estimated)

PRIMARY OUTCOMES:
LTVV Compliance | through study completion - 6 months
  Defined as: % of time each patient is on a compliant tidal volume for the duration of mechanical ventilation.
  Measured as: VC, PRVC, or VC+ with volume set to 6.5 ml/kg or less for each patient (proportion of mechanically ventilated hours, excluding hours on appropriate CPAP/PS)

SECONDARY OUTCOMES:
PEEP FI02 Compliance (continuous variable) | through study completion - 6 months
  Defined as: % of time each patient is on a compliant FI02 and PEEP combination.
  Measured as: using recommended (per most recently run oxygenation protocol) PEEP-FIO2 combinations, (proportion of ventilated hours, excluding the first four hours of mechanical ventilation and excluding hours on appropriate CPAP/PS)
Utilization of Ventilation Protocol (continuous) | through study completion - 6 months
  Defined as: % of time each patient is managed with the computerized ventilation protocol.
  Measured as: Running the computerized ventilation protocol whenever a ventilator check is performed and an arterial blood gas was done within the previous hour, excluding hours on appropriate CPAP/PS
Utilization of Oxygenation Protocol (continuous) | through study completion - 6 months
  Defined as: % of time each patient is managed with the computerized oxygenation protocol.
  Measured as: Running the computerized oxygenation protocol at least every four hours when a ventilator check was performed, excluding hours on appropriate CPAP/PS
LTVV Compliance >90% (binary) | through study completion - 6 months
  Defined as: meeting, or not meeting, the target LTVV compliance of >90% for each patient.
  Measured as: VC, PRVC, or VC+ with volume set to 6.5 ml/kg or less for 90% or more of mechanically ventilated hours, excluding hours on appropriate CPAP/PS
PEEP FI02 Compliance >70% (binary) | through study completion - 6 months
  Defined as: meeting, or not meeting, the target PEEP FI02 compliance of >70% for each patient.
  Measured as: Using recommended (per most recently run oxygenation protocol) PEEP-FIO2 combinations for at least 70% of mechanically ventilated hours (excluding the first four hours of mechanical ventilation and excluding hours on appropriate CPAP/PS)
Ventilator-Free Days (VFD) to Day 28 | through study completion - 6 months
% of Patients who do not survive to day 28 | through study completion - 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States

REFERENCES:
- [Derived] Peltan ID, Knighton AJ, Barney BJ, Wolfe D, Jacobs JR, Klippel C, Allen L, Lanspa MJ, Leither LM, Brown SM, Srivastava R, Grissom CK. Delivery of Lung-protective Ventilation for Acute Respiratory Distress Syndrome: A Hybrid Implementation-Effectiveness Trial. Ann Am Thorac Soc. 2023 Mar;20(3):424-432. doi: 10.1513/AnnalsATS.202207-626OC. PMID 36350983